CLINICAL TRIAL: NCT01248325
Title: Clinical Trial Unicenter, Phase III, Randomized, Double-blind, Comparative to Evaluate the Efficacy, Tolerability and Superiority of Luffa Operculate Nasal Solution 5mg/mL Compared With Saline Solution in the Relief of Nasal Obstruction.
Brief Title: A Study of Luffa Operculate Nasal Solution 5mg/mL Compared With Saline (NaCl 09%) for the Relief of Nasal Obstruction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zurita Laboratorio Farmaceutico Ltda. (Industry)
Responsible Party: Maria Pilar Michielin Zurita, Zurita Laboratório Farmacêutico Ltda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZUR-LO-2009
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Rhinitis; Sinusitis
MeSH Terms: conditions — Rhinitis; Sinusitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Luffa Operculate Nasal Solution 5mg/mL (Experimental): The treatment will start on the first visit in which subjects will be instructed to instill in the nasal passages, 3 drops of the product by morning and 3 drops of the product at night.
  Interventions: Drug: Luffa Operculate Nasal Solution 5mg/mL
- Saline Solution (NaCl 0,9%) (Active Comparator): The treatment will start on the first visit in which subjects will be instructed to instill in the nasal passages, 3 drops of the product by morning and 3 drops of the product at night.
  Interventions: Drug: Saline Solution (NaCl 0,9%)

INTERVENTIONS:
Drug: Luffa Operculate Nasal Solution 5mg/mL — The treatment will start on the first visit in which subjects will be instructed to instill in the nasal passages, 3 drops of the product by morning and 3 drops of the product at night.
  Arms: Luffa Operculate Nasal Solution 5mg/mL
Drug: Saline Solution (NaCl 0,9%) — The treatment will start on the first visit in which subjects will be instructed to instill in the nasal passages, 3 drops of the product by morning and 3 drops of the product at night.
  Arms: Saline Solution (NaCl 0,9%)

SUMMARY:
Sixty subjects will take part in this study. The subjects will be randomly assigned in a 1:1 ratio between the two arms of study. (Group A: Solution of Luffa Nasal Operculate 5mg/mL, Group B: saline).

The subjects will use the study medication or comparative, according to their randomization, for a treatment period of 3 to 7 days. A follow-up visit will be made 15 days after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged over 18 years.
* Presence of nasal congestion due to colds, rhinitis, influenza, sinusitis and acute or chronic sinusitis
* Sign the Informed Consent Form
* Comply the study requirements and attend to study visits
* Female subjects must have a NEGATIVE urine pregnancy test during the screening.

Exclusion Criteria:

* Known allergy to any study product component
* Subject pregnant, lactating or of childbearing potential and not using adequate and effective contraceptive
* Vasoconstrictor nasal topic or oral
* Use of a decongestant nasal whatever the route of administration
* Use of intranasal corticosteroids
* Use of antiallergic
* Use of medication containing atropine
* Subjects that are participating in another study or who participated in another study, less than 12 months
* Any subjects deemed unsuitable for study by the Principal Investigator
* Abuse of alcohol or illicit drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of nasal congestion | 3 days
  If the patient present a improvement of nasal congestion 3 days after the treatment start, the treatment will be discontinued and the patient will perfomr the Visit 2.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Gregório, doctor's, Principal Investigator — Universidade Federal de São Paulo/Hospital São Paulo/Escola Paulista de Medicina/UNIFESP
Locations (1):
- Universidade Federal de São Paulo/Hospital São Paulo/Escola Paulista de Medicina/UNIFESP, São Paulo, São Paulo, Brazil